CLINICAL TRIAL: NCT05837325
Title: Is the AMH Intrafollicular Level a Predictor of the Ploidy Status of the Blastocyst? A Prospective Study
Brief Title: Is the AMH Intrafollicular Level a Predictor of the Ploidy Status of the Blastocyst?
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2212-ABU-015-LM
Record Dates: First submitted 2023-03-13; First posted 2023-05-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Infertility, Female; Infertility
Keywords: Estradiol; FSH; LH; AMH; Ploidy; Chromosomes; Infertility; Progesterone; Inhibin B
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Sperm Injections, Intracytoplasmic; Culture Techniques; Biopsy; Vitrification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Follicular fluid Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Group
  Interventions: Procedure: ICSI; Procedure: Culture; Genetic: Biopsy; Procedure: Vitrification; Procedure: OPU - Study Group; Procedure: Denudation - Study Group
- Out of Study Group
  Interventions: Procedure: Oocyte Pick Up - Out of Study; Procedure: Denudation - Out of Study; Procedure: ICSI; Procedure: Culture; Genetic: Biopsy; Procedure: Vitrification

INTERVENTIONS:
Procedure: Oocyte Pick Up - Out of Study — Aspiration of follicles. search for the oocyte(s) All oocytes are grouped in one dish.
  Groups: Out of Study Group
Procedure: Denudation - Out of Study — All oocytes are denuded together. Maturational stages are recorded.
  Groups: Out of Study Group
Procedure: ICSI — One oocyte injected at a time.
Procedure: Culture — One embryo per culture drop. Individual follow-up of the embryo development.
Genetic: Biopsy — One embryo per culture drop.
Procedure: Vitrification — One embryo per vitrification straw.
Procedure: OPU - Study Group — Measure the size of the follicle and aspirate only one follicle and flush. The needle before moving to the second ovary. Oocyte included in the study will be cultured separately (each ovary separately too).
  Groups: Study Group
Procedure: Denudation - Study Group — Oocyte included in the study will be denuded separately. Maturational stages are recorded per follicle.
  Groups: Study Group

SUMMARY:
To investigate, whether on the day of egg retrieval, after ovarian stimulation for ICSI (intracytoplasmic sperm injection), there is a correlation between the intrafollicular AMH (Anti-Müllerian hormone) levels and the ploidy status of the blastocyst.

DETAILED DESCRIPTION:
In clinical practice, AMH is used as a diagnostic and/or prognostic marker in women in association with ovulation induction and in various pathophysiological conditions. This study looks to investigate if the hormonal environment that surrounds an oocyte has an impact on the ploidy status of the blastocyst. Nowadays, using NGS (Next Generation Sequencing) platform for analysis of 23 pairs of chromosomes for Preimplantation Genetic Testing on blastocysts, the ploidy status of the embryo is more adequately assessed. Furthermore, embryo culture to blastocyst will provide further information about embryo quality and possibilities of implantation.

To have complete information between the serum hormones, follicular hormones, embryo development and ploidy will provide to clinicians, embryologist and patients further information on embryo selection and adequate ovarian stimulation protocols.

The database will be exported from the clinical information manager, VRepro, to a table in excel format through a database-based query system. The exported data will be duly codified to protect the clinical and personal information of the participants. Prior to the statistical study, an exploratory data analysis will be carried out to review the quality of the information extracted.

ELIGIBILITY:
Inclusion Criteria:

* At least one follicle from each ovary at day of trigger
* Age from 18 to 40 years old
* Normal menstrual cycle of 25-35 days
* Poor, normal and high response will be included
* First follicle punctured from each ovary will be consider for inclusion: if the COC (Cumulus Oocyte Complex) is present in clear FF (Follicular fluid), the FF will be collected separately for further analysis and the oocyte included in the study

Exclusion Criteria:

* Very hematic follicular fluid
* If the COC is not found in the follicular fluid
* Azoospermia
* Known chromosomal abnormalities
* Severe OAT (Oligoasthenoteratozoospermia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Female undergoing IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oocyte maturity | 1 day
  Calculated as percentage transformation of an oocyte from prophase I to metaphase II
Fertilization | 1 day
  Percentage of mature oocytes - metaphase II (MII) that become 2 pronucleii embryos (2PN)
Blastulation | 1 day
  Ability of the embryo to form a cavity (=to blastulate) 114-118 hours post ICSI. Number of blastocysts divided by the number of 2PN
Blastocyst quality | 6 days
  Four Embryo Quality Scores (EQ1, 2, 3, 4) based on the expansion stage of the blastocyst, the grade of the inner cell mass and the grade of the trophectoderm.
Ploidy status | 14 days
  Determined after biopsy of trophectoderm cells, taken from the blastocyst on day 5, 6 or 7 from development
Mitochondria status | 14 days
  Measured as mtDNA ratio, the ratio of mitochondrial DNA (mtDNA) read counts to autosomal (chromosome 1-22) DNA read counts

SECONDARY OUTCOMES:
AMH in the follicular fluid. | 1 day
  To evaluate if there is an association between the levels of serum AMH on day 2-3 of the stimulation, AMH day of OPU and the intra-follicular AMH.
FSH in the follicular fluid. | 1 day
  To evaluate if there is an association between serum FSH on day 2-3 of the stimulation, serum FSH day of OPU and the intra-follicular FSH.
LH in the follicular fluid. | 1 day
  To evaluate if there is an association between serum LH on day 2-3 of the stimulation, serum LH day of OPU and the intra-follicular LH.
E2 in the follicular fluid. | 1 day
  To evaluate if there is an association between serum E2 on day 2-3 of the stimulation, serum E2 day of OPU and the intra-follicular E2.
P4 in the follicular fluid. | 1 day
  To evaluate if there is an association between serum P4 on day 2-3 of the stimulation, serum P4 day of OPU and the intra-follicular P4.
Inhibin B in the follicular fluid. | 1 day
  To evaluate if there is an association between serum Inhibin B on day 2-3 of the stimulation, serum Inhibin B day of OPU and the intra-follicular Inhibin B.
AMH in serum day of OPU | 1 day
  To evaluate if there is an association between the levels of serum AMH on day 2-3 of the stimulation, AMH day of OPU and the intra-follicular AMH.
FSH in serum day of OPU | 1 day
  To evaluate if there is an association between serum FSH on day 2-3 of the stimulation, serum FSH day of OPU and the intra-follicular FSH.
LH in serum day of OPU | 1 day
  To evaluate if there is an association between serum LH on day 2-3 of the stimulation, serum LH day of OPU and the intra-follicular LH.
E2 in serum day of OPU | 1 day
  To evaluate if there is an association between serum E2 on day 2-3 of the stimulation, serum E2 day of OPU and the intra-follicular E2.
P4 in serum day of OPU | 1 day
  To evaluate if there is an association between serum P4 on day 2-3 of the stimulation, serum P4 day of OPU and the intra-follicular P4.
Inhibin B in serum day of OPU | 1 day
  To evaluate if there is an association between serum Inhibin B on day 2-3 of the stimulation, serum Inhibin B day of OPU and the intra-follicular Inhibin B.
AMH in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between the levels of serum AMH on day 2-3 of the stimulation, AMH day of OPU and the intra-follicular AMH.
FSH in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between serum FSH on day 2-3 of the stimulation, serum FSH day of OPU and the intra-follicular FSH.
LH in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between serum LH on day 2-3 of the stimulation, serum LH day of OPU and the intra-follicular LH.
E2 in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between serum E2 on day 2-3 of the stimulation, serum E2 day of OPU and the intra-follicular E2.
P4 in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between serum P4 on day 2-3 of the stimulation, serum P4 day of OPU and the intra-follicular P4.
Inhibin B in serum day of day 2/3 of stimulation. | 1 day
  To evaluate if there is an association between serum Inhibin B on day 2-3 of the stimulation, serum Inhibin B day of OPU and the intra-follicular Inhibin B.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Melado, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hattori Y, Sato T, Okada H, Saito C, Sugiura-Ogasawara M. Comparison of follicular fluid and serum anti-Mullerian hormone levels as predictors of the outcome of assisted reproductive treatment. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(2):252-6. doi: 10.1016/j.ejogrb.2013.03.021. Epub 2013 Apr 25. PMID 23622971
- [Background] Capkin SI, Ozyer S, Karayalcin R, Moraloglu O, Ozcan S, Ugur M. Serum and follicular fluid Anti-Mullerian hormone concentrations at the time of follicle puncture and reproductive outcome. J Turk Ger Gynecol Assoc. 2012 Mar 1;13(1):21-6. doi: 10.5152/jtgga.2011.71. eCollection 2012. PMID 24627670
- [Background] Melado Vidales L, Fernandez-Nistal A, Martinez Fernandez V, Verdu Merino V, Bruna Catalan I, Bajo Arenas JM. Anti-Mullerian hormone levels to predict oocyte maturity and embryo quality during controlled ovarian hyperstimulation. Minerva Ginecol. 2017 Jun;69(3):225-232. doi: 10.23736/S0026-4784.16.03958-7. Epub 2016 Jun 28. PMID 27352270
- [Background] Hammoud I, Vialard F, Bergere M, Albert M, Gomes DM, Adler M, Malagrida L, Bailly M, Wainer R, Selva J. Follicular fluid protein content (FSH, LH, PG4, E2 and AMH) and polar body aneuploidy. J Assist Reprod Genet. 2012 Oct;29(10):1123-34. doi: 10.1007/s10815-012-9841-8. Epub 2012 Aug 14. PMID 22890422
- [Background] Calzada M, Lopez N, Noguera JA, Mendiola J, Hernandez AI, Corbalan S, Sanchez M, Torres AM. AMH in combination with SHBG for the diagnosis of polycystic ovary syndrome. J Obstet Gynaecol. 2019 Nov;39(8):1130-1136. doi: 10.1080/01443615.2019.1587604. Epub 2019 Jun 17. PMID 31208261
- [Background] Devroey P, Aboulghar M, Garcia-Velasco J, Griesinger G, Humaidan P, Kolibianakis E, Ledger W, Tomas C, Fauser BC. Improving the patient's experience of IVF/ICSI: a proposal for an ovarian stimulation protocol with GnRH antagonist co-treatment. Hum Reprod. 2009 Apr;24(4):764-74. doi: 10.1093/humrep/den468. Epub 2009 Jan 19. PMID 19153090
- [Background] Ferraretti AP, Gianaroli L. The Bologna criteria for the definition of poor ovarian responders: is there a need for revision? Hum Reprod. 2014 Sep;29(9):1842-5. doi: 10.1093/humrep/deu139. Epub 2014 Jul 9. PMID 25008235